CLINICAL TRIAL: NCT00555087
Title: Treatment of Erectile Dysfunction in Hypogonadal Men With Testosterone Undecanoate i.m. 1000 mg. A Prospective, Multi-Center Clinical Study Phase IV.
Brief Title: Treatment of Erectile Dysfunction in Hypogonadal Men With Testosterone Undecanoate
Acronym: Nebidolocal
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Santa Fe (Other)
Collaborators: Bayer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/1084
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Erectile Dysfunction; Hypogonadotrophic Males
Keywords: Erectile dysfunction; Hypogonadotrophic males
MeSH Terms: conditions — Erectile Dysfunction | interventions — testosterone undecanoate; Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A= Nebido (Experimental): It is and intervention study with 1 arm
  Interventions: Drug: Testosterone Undecanoate and/or PDE-5

INTERVENTIONS:
Drug: Testosterone Undecanoate and/or PDE-5 — Testosterone Undecanoate 1000 mg IM injection; PDF5 tab, 20 mg
  Other Names: Nebido; Levitra

SUMMARY:
The main objective of this study is to evaluate the response of erectile dysfunction in hypogonadotrophic males with Testosterone undecanoate i.m. as per IIEF and the question of the GAQ (Global Evaluation Questionnaire) after 42 weeks of treatment.

Secondary Study Objectives

* To monitor adverse events and changes in hemoglobin and serum chemistry with: PSA, lipid profile, renal-hepatic profile and glycemia, and control by means of a rectal digital examination.
* To Determinate physiologic reconstitution in patients under treatment by means of total and free testosterone dosage.

DETAILED DESCRIPTION:
The importance of testosterone in desire, interest and sexual motivation is well known, but its effects on erectile function continue provoking controversy. Data obtained in animals under experimental or surgical castration, explains how this condition can cause a veno-occlusive dysfunction and therefore an erectile dysfunction. In a model of animal flebogenous erectile dysfunction, the intracavernous vascular endothelial growth factor (VEGF), together with testosterone, reestablishes the balance between the muscle and the conjunctive tissue, hypertrophy and hyperplasia of endothelial cells and regularizes the diameter of dorsal nervous cells, thus preventing the veno-occlusive dysfunction. Castration also induces the apopthosis in the erectile tissue of the penis; the treatment with testosterone provokes a new DNA synthesis.

There are certain indicators that the treatment with testosterone could help patients with erectile dysfunction and low testosterone base line amounts. Likewise, androgens could control the expression and the activity of type 5 phosphodiesterase (PDE-5) of the cavernous body of the penis.

Pharmacological treatment with PDE-5 inhibitors, administered orally fails in certain cases of erectile dysfunction, even more in hypogonadal males. Some studies show that the combination of testosterone with a PDE-5 inhibitor helps the recovery of sexual function in patients; therefore, giving the possibility of a combined pharmacological treatment with testosterone in erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old and younger than 70 years.
* To have diagnosis of erectile dysfunction by IIEF. Qualification less than 46 points and/or GAQ with Answer "NO".
* Patients with Inform consent letter signed.
* Patients without any therapy with other type of testosterone, gonadotrophines and/or PDE-5 in the previous 4 weeks of their inclusion at the study.
* Diagnosis of hypogonadism according to the criteria:
* Testosterone dosage lower than 12 nmol/L
* Free testosterone shall be below 180 pmol/L o 52 pg/mL

Exclusion Criteria:

* People less than 18 years old and older than 70 years.
* Patients with history of or with known or suspected sleep apnea.
* Patients who participate in other study protocols
* Known or suspected active systemic infection.
* Patients with HIV + and/ or known HTLV+.
* Patients with hyperprolactinemia
* Patients with known or suspected coagulopathies
* Patients with Klinefelter
* Known or suspected psychiatric illness.
* Patients who have received prior therapy with some kind of testosterone in the last 4 months or a PDE-5 inhibitor in the last month.
* Patients with contraindications for the use of PDE-5 inhibitors
* Patients having a diagnosis of erectile dysfunction but with total and/ or free testosterone levels within the physiological range.
* Patients with APE ≥ 2.5 ng/ml in younger than 60 years, or > de 3 ng/ml in older than 60 years.
* Abnormal prostate findings during the digital rectal examination (that is to say, irregularities, hard consistency when examined).
* Concomitant malignant diseases or history of prostate cancer

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-05; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Score higher than or equal to 21 of the erectile dysfunction domain of the IIEF, or response to treatment | 42 weeks
and/or an affirmative response to the GAQ will be considered for the analysis | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Jaspersen, MD, Principal Investigator — H Santa Fe
Locations (3):
- Mexico (3):
  - Hospital Santa Fe, Mexico City, D.F.
  - Hospital General de Occidente, Guadalajara, Jalisco
  - Hospital Universitario de Nuevo León, Monterrey, Nuevo León